CLINICAL TRIAL: NCT00920582
Title: A Phase 3, Randomized, Double-Blind, Multinational, Placebo-Controlled Study to Evaluate Efficacy and Safety of Teplizumab (MGA031), a Humanized, FcR Non-Binding, Anti-CD3 Monoclonal Antibody, in Children and Adults With Recent-Onset Type 1 Diabetes Mellitus
Brief Title: Protege Encore Study- Clinical Trial of Teplizumab (MGA031) in Children and Adults With Recent-Onset Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: MacroGenics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-MGA031-03
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Herold Regimen (Experimental): 14-day cycle of teplizumab consisting of daily IV doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, and 413 µg/m2 on Study Days 1-4, respectively, and one dose of 826 µg/m2 on each of Study Days 5-14. Repeat at Week 26
  Interventions: Biological: Teplizumab Herold Regimen
- 33.3% Herold Regimen (Experimental): Subjects received a 14-day cycle of teplizumab consisting of daily IV doses of 17 µg/m2, 34 µg/m2, 68 µg/m2, and 136 µg/m2 on Study Days 1-4, respectively, and one dose of 273 µg/m2 on each of Study Days 5-14. Repeat at Week 26
  Interventions: Biological: Teplizumab 33.3% Herold Regimen
- Curtailed Herold Regimen (Experimental): Subjects received a 6 day cycle of teplizumab consisting of daily IV doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, and 413 µg/m2 on Study Days 1-4, respectively, and one dose of 826 µg/m2 on each of Study Days 5-6, followed by 8 days of IV placebo (Study Days 7-14). Repeat at Week 26
  Interventions: Biological: Teplizumab Curtailed Herold Regimen
- Placebo (Placebo Comparator): 14-day cycle of placebo consisting of daily IV doses. Repeat at Week 26
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Teplizumab Herold Regimen — Full dose of teplizumab IV for 14 days, repeated at Week 26
  Other Names: MGA031
  Arms: Herold Regimen
Drug: Placebo — IV dosing daily for 14 days repeated at Week 26
  Arms: Placebo
Biological: Teplizumab 33.3% Herold Regimen — One third full dose of teplizumab IV for 14 days, repeated at Week 26
  Other Names: MGA031
  Arms: 33.3% Herold Regimen
Biological: Teplizumab Curtailed Herold Regimen — Full dose of teplizumab IV for 6 days followed by placebo for 8 days, repeated at Week 26
  Arms: Curtailed Herold Regimen

SUMMARY:
The primary purpose of this study is to determine whether teplizumab (MGA031) infusions lead to greater reductions in insulin requirements in conjunction with near normal blood sugar control compared to placebo in patients recently diagnosed with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 8-35 years old
2. Body weight > 36 Kg
3. Diagnosis of diabetes mellitus according to the American Diabetes Association (ADA) criteria
4. Randomization on Study Day 0 within 12 weeks of first visit to any physician for symptoms or signs of diabetes
5. Requires insulin for T1DM or has required insulin at some time between diagnosis and administration of study drug
6. Detectable fasting or stimulated C-peptide level (above the lower limit of the reportable range of the assay) at screening
7. Diagnosis of T1DM as evidenced by one positive result on testing for any of the following antibodies at screening:

   * Islet-cell autoantibodies 512 (ICA512)/islet antigen-2 (IA-2),
   * Glutamic acid decarboxylase (GAD) autoantibodies, or
   * Insulin autoantibodies (in subjects on insulin for more than 2 weeks, ICA512/IA-2 or GAD must be positive).

Exclusion Criteria:

1. Prior administration of a monoclonal antibody-within the 1 year before randomization
2. Participation in any type of therapeutic drug or vaccine clinical trial within the last 12 weeks before randomization at Study Day 0
3. Any medical condition that, in the opinion of the investigator, would interfere with safe completion of the trial
4. Pregnant females or lactating females who intend to provide their own breast milk to the baby during the study
5. Current therapy with GLP-1 receptor agonists (e.g., exenatide or pramlintide), or any other agents that might stimulate pancreatic beta cell regeneration or insulin secretion
6. Current treatment with oral antidiabetic agents
7. Evidence of active or latent tuberculosis
8. Vaccination with a live virus or organism within the 8 weeks before randomization continuing through Week 52 of the study.

   * Influenza vaccination with a killed virus, including booster vaccinations, within 4 weeks before or after each dosing cycle.
   * Vaccination with other antigens or killed organisms within 8 weeks before or after each dosing cycle
9. Any infectious mononucleosis-like illness within the 6 months before randomization

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 254 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (118):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - NEA Clinic, Jonesboro, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Clinical Innovations Inc. Research Facility, Costa Mesa, California
  - Axis Clinical Trials, Los Angeles, California
  - Diabetes Associates Medical Group, Inc, Orange, California
  - Clinical Innovations, Inc., Riverside, California
  - San Diego Clinical Trials, San Diego, California
  - Ronald Chochinov Md Inc, Ventura, California
  - Yale University, New Haven, Connecticut
  - Christiana Care Research Institute, Newark, Delaware
  - Richard Hays, MD, Wellington, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - John H Stoger Jr. Hospital of Cook County, Cook County Hospital, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Mid-America Diabetes Associates, Wichita, Kansas
  - St. Agnes Hospital, Baltimore, Maryland
  - Maryland Diabetes & Endocrine Associates, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Alzohaili Medical Consultants, Dearborn, Michigan
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - University of Missouri - Columbia, Cosmopolitan Diabetes and Endocrinology, Columbia, Missouri
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Albany Medical College, Albany, New York
  - Bassett Healthcare, Cooperstown, New York
  - East Carolina University, Brody School of Medicine, Greenville, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - GHS Pediatric Endocrinology, Greenville, South Carolina
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Houston Center for Clinical Research, Houston, Texas
  - Medical & Surgical Clinic of Irving, Irving, Texas
  - InVisions Consultants, LLC, San Antonio, Texas
  - Diabetes and Glandular Disease Research Associates, PA, San Antonio, Texas
  - Endocrine Research Specialists, Ogden, Utah
  - Virginia Commonwealth University-Division of Pediatric Endocrinology & Metabolism, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerp
  - Cliniques du Sud Luxembourg - Vivalia, Arlon
- Czechia (5):
  - I. Detska interni klinika,Fakultni nemocnice Brno Detska nemocnice, Brno
  - Klinika deti a dorostu FN Kralovske Vinohrady, Prague
  - Centrum diabetologie, Institut klinicke a experimentalni mediciny, Prague
  - Pediatricka klinika UK 2.LF a FN Motol, Fakultni nemocnice v Motole, Prague
  - Detska klinika, Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Central Hospital of Mikkeli, Mikkeli
  - Oulu University Hospital, Oulu
- France (6):
  - CHU de Besançon, Besançon
  - CHU de Brest Hôpital de la Cavale Blanche, Brest
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU de Bordeaux, Pessac
  - CHU de Reims, Reims
  - Hôpitaux Universitaires de Strasbourg Hôpital Civil, Strasbourg
- Germany (8):
  - Diabetes-Klinik Bad Nauheim GmbH, Bad Nauheim
  - Herz und Diabeteszentrum Nordrhein-Westfallen, Bad Oeynhausen
  - Charite, Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitatsklinik Giessen, Giessen
  - Asklepios Westklinikum Hamburg, Hamburg
  - Kinderkrankenhaus auf der Bult, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
- India (16):
  - Medwin Hospitals, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - DHL Research Centre, Ahmedabad, Gujarat
  - Bangalore Diabetes Centre, Bangalore, Karnataka
  - Health & Research Centre, Trivandrum, Kerala
  - Gandhi's Research Institute, Nagpur, Maharashtra
  - Grant Medical Foundation, Pune, Maharashtra
  - KEM Hospital Research Center, Pune, Maharashtra
  - Maulana Azad Medical College and Associated Hospitals, New Delhi, National Capital Territory of Delhi
  - Kalinga Hospital Limited, Bhubaneswar, Odisha
  - Diabetes-Thyroid-Hormone Research Institute Pvt. Ltd., Madhya, Pradesh
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - Fortis Escorts Hospital, Jaipur, Rajasthan
  - Hormone Care & Research Center, Ghaziabad, Uttar Pradesh
  - B. P. Poddar Hospital & Medical Research Limited, Kolkata, West Bengal
  - Apollo Glenagles Hospital, Kolkata, West Bengal
- Israel (5):
  - Hillel Yaffe Medical Center, Hadera
  - Mayer Children's Hospital of Haifa, Haifa
  - The E. Wolfson Medical Center, Holon
  - Schneider Children's Medical, Petah Tikva
  - The Safra Children's Hospital, The Chaim Sheba Medical Center, Ramat Gan
- Italy (3):
  - Struttura Complessa di Pediatria, Azienda Ospedaliero-Universitaria di Modena,, Modena
  - U.O. di Malattie del Metabolismo, Pisa
  - U.O. di Malattie Metaboliche e Diabetologia, Pisa
- Mexico (3):
  - Hospital y Clinica OCA / Monterrey International Research Center, Monterrey, Nuevo León
  - Medical Care & Research, Mérida, Yucatán
  - Centro Especializado en Diabetes, Obesidad y Prevención de Enfermedades Cardiovasculares, S.C., Mexico City
- Stichting Diabeter, Rotterdam, Netherlands
- Poland (6):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wojewódzki Specjalistyczny Szpital Dzieciecy, Kielce
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Uniwersytecki Szpital Kliniczny Nr 4, Lodz
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny w Warszawie-Filia, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr1 we Wroclawiu, Wroclaw
- Romania (3):
  - S.C. Minimed S.R.L., Bacau
  - Institutul National De Diabet, Nutritie si Boli Metabolice, Bucharest
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare
- Spain (2):
  - Hospital Universitario Principe de Asturias, Alcalá de Henares
  - Hospital Dr. Josep Trueta, Girona
- Ukraine (7):
  - Donetsk Regional Children Clinical Hospital, Donetsk
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Ivano-Frankivsk State Regional Pediatric Clinical Hospital, Ivano-Frankivsk
  - Kharkiv Regional Clinical Children Hospital, Department of Endocrinology, Kharkiv
  - Ukrainian Children Specialized Clinical Hospital, Kyiv
  - Institute of Endocrinology and Metabolism named after V.Komisarenko of AMS Ukraine, Kyiv
  - Regional Clinical Endocrinology Dispensary of MoH Ukraine, Vinnitsa
- United Kingdom (6):
  - George Eliot Hospital NHS Trust, Nuneaton, Warwickshire
  - University of Bristol Henery Wellcome laboratories for Integrative Neuroscience and Endocrinology,, Bristol
  - Aintree University Hospitals NHS Foundation Trust, Liverpool
  - Kings College, Clinical Research Unit, Department of Diabetes and Endocrinology, London
  - Queens Medical Centre, Diabetes and Endocrinology Unit, Nottingham
  - Sheffield Children's Hospital NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Started | 63 | 66 | 63 | 62
Completed | 50 | 60 | 52 | 57
Not Completed | 13 | 6 | 11 | 5
Not completed — Lost to Follow-up | 5 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 6 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo | Total
Number analyzed (Participants) | 63 | 66 | 63 | 62 | 254
Age, Continuous [Median (Full Range); unit: years] | 16.0 [8.0 to 23.0] | 16.0 [8.0 to 35.0] | 15.0 [8.0 to 33.0] | 16.0 [9.0 to 35.0] | 16.0 [8.0 to 35.0]
Age, Customized [Count of Participants; unit: Participants]
  8-11 years | 13 | 12 | 13 | 11 | 49
  12-17 years | 24 | 29 | 24 | 25 | 102
  18-35 years | 26 | 25 | 26 | 26 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 17 | 21 | 83
  Male | 38 | 46 | 46 | 41 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 4 | 6
  Not Hispanic or Latino | 63 | 65 | 62 | 58 | 248
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 25 | 26 | 25 | 23 | 99
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 2 | 5
  White | 36 | 39 | 35 | 37 | 147
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Romania | 3 | 3 | 1 | 3 | 10
  United States | 17 | 17 | 17 | 17 | 68
  Czechia | 4 | 5 | 6 | 5 | 20
  Ukraine | 5 | 5 | 4 | 6 | 20
  United Kingdom | 0 | 0 | 1 | 0 | 1
  India | 25 | 26 | 25 | 23 | 99
  Spain | 1 | 2 | 2 | 2 | 7
  Belgium | 1 | 0 | 0 | 0 | 1
  Finland | 0 | 1 | 0 | 0 | 1
  Poland | 3 | 2 | 2 | 2 | 9
  Mexico | 0 | 0 | 0 | 1 | 1
  Israel | 3 | 3 | 4 | 2 | 12
  Germany | 1 | 2 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and Hemoglobin A1c (HbA1c) Level of Less Than 6.5%.
Time Frame: 52 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 63 | 66 | 63 | 62
Participants | 8 | 8 | 9 | 6
Statistical Analysis 1: Comparison: Herold Regimen vs Placebo; Test type: Superiority; p = 0.609, Mantel Haenszel; Odds Ratio (OR) = 1.348, 95% CI 2-sided [0.431 to 4.219]
Statistical Analysis 2: Comparison: 33.3% Herold Regimen vs Placebo; Test type: Superiority; p = 0.601, Mantel Haenszel; Odds Ratio (OR) = 1.356, 95% CI 2-sided [0.453 to 4.230]
Statistical Analysis 3: Comparison: Curtailed Herold Regimen vs Placebo; Test type: Superiority; p = 0.400, Mantel Haenszel; Odds Ratio (OR) = 1.624, 95% CI 2-sided [0.521 to 5.066]

2. Primary Outcome: Mean Change From Baseline in HbA1c Between Teplizumab and Placebo
Time Frame: 52 weeks after randomization
Population: Analysis population includes all participants with available data at 52 weeks after randomization.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 54 | 59 | 54 | 58
percent HbA1c | 0.01 (1.803) | -0.02 (2.169) | 0.35 (25.12) | 0.03 (2.566)

3. Secondary Outcome: The Change in Beta-cell Function as Measured by C-peptide Secretory Response Following a Mixed Meal
Time Frame: 52 weeks after randomization
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 29 | 30 | 27 | 26
nmol/L | 0.04 (0.276) | -0.05 (0.456) | 0.04 (0.287) | -0.04 (0.419)
Statistical Analysis 1: Comparison: Herold Regimen vs Placebo; Test type: Superiority; p = 0.365, ANCOVA; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.086 to 0.031]
Statistical Analysis 2: Comparison: 33.3% Herold Regimen vs Placebo; Test type: Superiority; p = 0.842, ANCOVA; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.078 to 0.064]
Statistical Analysis 3: Comparison: Curtailed Herold Regimen vs Placebo; Test type: Superiority; p = 0.565, ANCOVA; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [-0.089 to 0.171]

4. Secondary Outcome: The Change in Beta-cell Function as Measured by C-peptide Secretory Response Following a Mixed Meal
Time Frame: 104 weeks after randomization
Population: The study was terminated early and no data for C-peptide secretory response following a mixed meal was collected at Week 104. Measurement of C-peptide response after a mixed meal at selected timepoints up to Week 104 was replaced with measurement of fasting C-peptide levels at Day 365 by protocol amendment. Data were collected only at Days 141 and 365, due to the early termination of the study.
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Mean Number of Total, Major, Minor and Nocturnal Hypoglycemia Events
Description: Number of hypoglycemic events by type per participant
Time Frame: Throughout the study up to 2 years
Population: Analysis of hypoglycemic events at 52 weeks and 104 weeks was combined in the statistical analysis plan. The presentation reflects the total hypoglycemic events throughout the study.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 63 | 66 | 63 | 62
events
  Total (any) | 13.7 (22.35) | 15.9 (22.90) | 18.9 (41.42) | 15.5 (22.70)
  Minor hypoglycemia | 4.1 (6.97) | 4.4 (6.38) | 5.4 (12.11) | 4.7 (10.45)
  Major hypoglycemia | 10.0 (0.13) | 0.1 (0.42) | 0.0 (0.18) | 0.0 (0.13)
  Nocturnal hypoglycemia | 2.0 (3.17) | 2.1 (5.54) | 1.4 (2.46) | 1.6 (3.33)

6. Secondary Outcome: Mean Number of Daily Insulin Injections
Time Frame: 52 weeks after randomization
Population: The number of daily insulin injections was not collected. Insulin use was analyzed as units/kg/day, not by number of injections.
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and Hemoglobin A1c (HbA1c) Level of Less Than 6.5%.
Time Frame: 104 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 14 | 13 | 15 | 17
Participants | 1 | 2 | 1 | 1

8. Secondary Outcome: The Proportion of Subjects Who Have Both a Total Daily Insulin Dose < 0.5 U/Kg/Day and Hemoglobin A1c (HbA1c) Level < 7.0%
Time Frame: 52 weeks after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 63 | 66 | 63 | 62
Participants | 13 | 10 | 12 | 7
Statistical Analysis 1: Comparison: Herold Regimen vs Placebo; Test type: Superiority; p = 0.142, Mantel Haenszel; Odds Ratio (OR) = 2.197, 95% CI 2-sided [0.764 to 6.312]
Statistical Analysis 2: Comparison: 33.3% Herold Regimen vs Placebo; Test type: Superiority; p = 0.460, Mantel Haenszel; Odds Ratio (OR) = 1.487, 95% CI 2-sided [0.517 to 4.278]
Statistical Analysis 3: Comparison: Curtailed Herold Regimen vs Placebo; Test type: Superiority; p = 0.199, Mantel Haenszel; Odds Ratio (OR) = 1.954, 95% CI 2-sided [0.690 to 5.532]

9. Secondary Outcome: The Mean HbA1c Change From Baseline
Time Frame: 104 weeks after randomization
Population: No statistical analysis was performed on the limited data collected at 104 weeks after randomization. Only descriptive statistics are provided.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 15 | 14 | 15 | 21
percent glycosylated hemoglobin | 1.05 (2.344) | 1.11 (2.494) | 0.71 (3.740) | 1.21 (2.857)

10. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: throughout the study, up to 104 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 63 | 66 | 63 | 62
Participants | 63 | 66 | 63 | 62

11. Secondary Outcome: Number of Participants With Serious Adverse Events
Time Frame: throughout the study, up to 104 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
Number analyzed (Participants) | 63 | 66 | 63 | 62
Participants | 7 | 6 | 8 | 3

ADVERSE EVENTS:
Time Frame: Throughout the study, up to 2 years
Description: All AEs and SAEs were reported from Day 0 to Day 364. Only treatment-related non-serious AEs, and all SAEs were reported after Day 364.
Arm/Group | Herold Regimen | 33.3% Herold Regimen | Curtailed Herold Regimen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/66 | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 7/63 | 6/66 | 8/63 | 3/62
Other Adverse Events (participants affected / at risk) | 63/63 | 66/66 | 63/63 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herold Regimen (N=63) | 33.3% Herold Regimen (N=66) | Curtailed Herold Regimen (N=63) | Placebo (N=62)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 — too few lymphocytes
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 1 | 0 | 0
Hepatic amoebiasis (Infections and infestations) | 0 | 0 | 1 | 0 — Entamoeba infection in the liver
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 — kidney infection
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 — stomach flu
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 — too much sugar, not enough insulin
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 — seizure from low blood sugar
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 — too much blood sugar
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — not enough blood sugar
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 — unconscious due to low blood sugar
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Herold Regimen (N=63) | 33.3% Herold Regimen (N=66) | Curtailed Herold Regimen (N=63) | Placebo (N=62)
Lymphopenia (Blood and lymphatic system disorders) | 26 | 21 | 25 | 6 — too few lymphocytes
Leukopenia (Blood and lymphatic system disorders) | 11 | 12 | 11 | 9 — too few white blood cells
Neutropenia (Blood and lymphatic system disorders) | 7 | 8 | 5 | 5 — too few blood neutrophils
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 7 — too few red blood cells
Nausea (Gastrointestinal disorders) | 6 | 5 | 4 | 7
Vomiting (Gastrointestinal disorders) | 3 | 3 | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 4 | 2
Pyrexia (General disorders) | 14 | 12 | 20 | 7 — fever
Chills (General disorders) | 5 | 2 | 5 | 4
Epstein-Barr viraemia (Infections and infestations) | 13 | 5 | 6 | 3 — Epstein-Barr Virus infection
Nasopharyngitis (Infections and infestations) | 3 | 8 | 8 | 5 — sore throat
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 6 | 6
Pharyngitis (Infections and infestations) | 3 | 1 | 2 | 5 — sore throat
Blood bicarbonate decreased (Investigations) | 31 | 38 | 27 | 26
Lymphocyte count decreased (Investigations) | 35 | 32 | 33 | 6
White blood cell count decreased (Investigations) | 39 | 28 | 29 | 13
Haemoglobin decreased (Investigations) | 23 | 20 | 22 | 17
Neutrophil count decreased (Investigations) | 23 | 16 | 23 | 10
Aspartate aminotransferase increased (Investigations) | 20 | 15 | 22 | 11
Alanine aminotransferase increased (Investigations) | 20 | 14 | 19 | 6
Blood potassium increased (Investigations) | 16 | 12 | 14 | 12
Blood sodium decreased (Investigations) | 9 | 17 | 14 | 16
Blood calcium decreased (Investigations) | 20 | 13 | 8 | 11
Platelet count decreased (Investigations) | 19 | 13 | 11 | 6
Blood alkaline phosphatase increased (Investigations) | 11 | 12 | 12 | 8
Blood calcium increased (Investigations) | 6 | 5 | 7 | 7
Blood bilirubin increased (Investigations) | 7 | 9 | 3 | 3
Epstein-Barr virus antibody positive (Investigations) | 6 | 6 | 4 | 6
Blood phosphorus increased (Investigations) | 5 | 6 | 6 | 2
Blood albumin decreased (Investigations) | 6 | 3 | 5 | 2
Blood creatinine increased (Investigations) | 4 | 4 | 5 | 2
Gamma-glutamyltransferase increased (Investigations) | 4 | 2 | 7 | 1
Blood sodium increased (Investigations) | 6 | 4 | 1 | 1
Eosinophil count increased (Investigations) | 3 | 3 | 4 | 1
Blood chloride decreased (Investigations) | 4 | 3 | 2 | 2
Blood potassium decreased (Investigations) | 5 | 2 | 3 | 0
Blood bicarbonate increased (Investigations) | 2 | 4 | 3 | 1
Red blood cell count decreased (Investigations) | 5 | 1 | 2 | 1
Bilirubin conjugated increased (Investigations) | 5 | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 6 | 10 | 13 — not enough sodium in the bloodstream
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 7 | 7 | 9 — not enough calcium in the bloodstream
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 8 | 8 | 5 — too much potassium in the bloodstream
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 6 | 2 — not enough sugar in the bloodstream
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 1 | 3 | 3 — not enough albumin in the bloodstream
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 5 | 1 — too much calcium in the bloodstream
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 5 | 1 — muscle pain
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0
Headache (Nervous system disorders) | 14 | 11 | 15 | 12
Depression (Psychiatric disorders) | 4 | 1 | 0 | 1
proteinuria (Renal and urinary disorders) | 4 | 7 | 3 | 5 — protein in the urine
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 5 | 1 — mouth and throat pain
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 9 | 9 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 9 | 8 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 7 | 4 | 4 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 7 | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 1 | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 0
urticaria (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1 — itchy rash
Fatigue (General disorders) | 1 | 3 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less